CLINICAL TRIAL: NCT03432195
Title: A Phase 1, Crossover Study to Evaluate the Pharmacokinetics of Corplex™ Donepezil 10 mg Transdermal Delivery System Applied to Different Body Locations
Brief Title: A Clinical Study to Evaluate the Pharmacokinetics (PK) of Corplex™ Donepezil Transdermal Delivery System (TDS) Applied to Different Body Locations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P16012
Record Dates: First submitted 2018-01-31; First posted 2018-02-14 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Donepezil TDS Back (Experimental): Corplex Donepezil TDS 10 mg/day applied to the Back for 1 week (7 days)
  Interventions: Drug: Donepezil TDS
- Donepezil TDS Buttock (Experimental): Corplex Donepezil TDS 10 mg/day applied to the Buttock for 1 week (7 days)
  Interventions: Drug: Donepezil TDS
- Donepezil TDS Leg (Experimental): Corplex Donepezil TDS 10 mg/day applied to the Leg for 1 week (7 days)
  Interventions: Drug: Donepezil TDS

INTERVENTIONS:
Drug: Donepezil TDS — Donepezil Hydrochloride Transdermal Delivery System

SUMMARY:
A Phase 1, Crossover Study to Evaluate the Pharmacokinetics of Corplex™ Donepezil 10 mg Transdermal Delivery System Applied to Different Body Locations

DETAILED DESCRIPTION:
Randomized, open-label, 3-way crossover study

Up to 66 healthy, adult male and female subjects will be enrolled.

All subjects will receive Corplex Donepezil TDS patches applied to 3 different locations on each subject (back, buttock, and leg) during 3 different, consecutive treatment periods. For each subject, the location of product administration during each treatment period will be randomized.

During each treatment period, all subjects will receive a once-weekly 10 mg TDS, target dose 10 mg donepezil/day, applied for 7 days (1 week) on either the back, buttock, or leg in accordance with the randomized treatment location for that treatment period.

Blood samples for donepezil PK will be collected pre-dose until the end of each treatment period. The PK sample collection time points are as follows:

Week 1: Pre-TDS application prior to 0 hour and post-TDS application at 2, 6, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, and 156 hours.

Week 2: Pre-Week 1 TDS removal at 168 hours, and post-TDS removal at up to 528 hours

Adhesion and skin irritation will be monitored throughout TDS treatments. Safety will be monitored throughout the study by adverse event reporting, repeated clinical and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female
* Body mass index ≥ 18.0 and ≤ 32.0 kg/m2 at screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), as deemed by the Investigator
* Have a Fitzpatrick skin type of I, II or III or have skin colorimeter scores equivalent to the allowed Fitzpatrick skin type

Key Exclusion Criteria:

* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds (including piperidine derivatives and other cholinesterase inhibitors)
* Has intolerance to venipuncture and/or inability to comply with the extensive blood sampling required for this study or does not have suitable veins in both arms
* Potential for occupational exposure to anticholinesterase agents
* Estimated creatinine clearance in non-elderly subjects <80 mL/min at screening and in elderly subjects (i.e., ≥55 years of age) <60 mL/min at screening
* Hemoglobin value of less than 11.5 g/dl for females, 13.0 g/dl for males at screening and first check-in
* Muscle relaxants, anti-Parkinsonian or neuroleptic medications prior to the first dose of study drug
* History or presence of significant skin damage or other skin disturbances as deemed by the Investigator to potentially interfere with patch procedures
* Use of donepezil hydrochloride or related drugs within 60 days prior to the first study drug administration
* Clinically significant depression symptoms or suicidal ideation or behavior as determined by the Investigator

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics, AUC | Blood samples for donepezil PK will be collected pre-dose until the end of each treatment period, approximately 18 weeks total
  Area under the plasma concentration versus time curve (AUC) of once-weekly Corplex Donepezil TDS applied to different body locations.
Pharmacokinetics, CMAX | Blood samples for donepezil PK will be collected pre-dose until the end of each treatment period, approximately 18 weeks total
  Peak Plasma Concentration (Cmax) of once-weekly Corplex Donepezil TDS applied to different body locations.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Daily during 1 week treatment period throughout the 5 week period
  General Safety (adverse events and serious adverse events as reported by subject following guidance CTCAE v4.0)
Summary Listing of Skin Irritation Score of Donepezil Corplex TDS by post-removal time point | 0.5hr, 24hr, 48hr and 72hr after each TDS removal. (3 days)
  Skin irritation score is determined by the sum of Dermal Response score (8-point categorical scale; where 0=no evidence of irritation to 7=strong reaction) using numeric values) and the Other Effects score (6-point categorical scale where 0=none observed to H=scabs/erosion using alphabet letters equivalent to numeric values) and summarized by application site (back, buttock and leg)
Application Site Mean Adhesion Scores of Donepezil Corplex TDS | Daily during 1 week treatment period
  Adhesion score is collected using a 12-point categorical scale, where 0=100% adhered to 11=detached

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
no plans